CLINICAL TRIAL: NCT06129071
Title: Analgesic Effect Evaluation of Ultrasound Guided Maxillary Nerve Block in Trigeminal Neuralgia
Brief Title: Analgesic Effect of Ultrasound Guided Maxillary Nerve Block in Trigeminal Neuralgia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: the principal investigator changed her mind and gave up from the study
Sponsor: Varazdin General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20061988
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-11

CONDITIONS: Trigeminal Neuralgia
Keywords: trigeminal neuralgia; maxillary nerve; ultrasound guided nerve block
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- US block of maxillar nerve (Experimental): Extraoral ultrasound-guided block of the maxillary nerve will be performed using an ultrasound device. After visualisation of the pterygomandibular space, of the maxillary artery and the mandibular nerve next to it, at a depth of 2-4 cm, the detection of the maxillary artery is confirmed by Color Doppler. A needle enters between the coronoid and condylar processes, using the "out of plane" technique, near the maxillary artery, and after negative aspiration, local anesthetic levobupivacaine (0,5%, 2 mL) combined with triamcinolonacetonid (2mL).
  Interventions: Procedure: US guided block of maxillary nerve

INTERVENTIONS:
Procedure: US guided block of maxillary nerve — Extraoral ultrasound-guided block of the maxillary nerve will be performed in the examined group using an ultrasound device and local anesthetic levobupivacaine (0,5%, 2 mL) combined with triamcinolonacetonid (2mL).

SUMMARY:
This is a study about the dynamics and effects of ultrasound guided maxillary nerve block in trigeminal neuralgia

DETAILED DESCRIPTION:
Standard pharmacological treatment for trigeminal neuralgia is often insufficient. In this setting, patients often suffer trough everyday activities and quality of life is disturbed substantially.

In this prospective clinical study, analgesic effect of ultrasound (US) guided maxillary nerve block will be investigated, in order to prolong pain-free time, reduce the use of standard analgesics, as well as atypical ones (e.g. antiepileptic drugs and antidepressants).

Characteristics of US guided maxillary nerve block will pain investigated: reduction of pain (decrease of VAS score), duration of pain-free period, pain level during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* patients with trigeminal neuralgia

Exclusion Criteria:

* allergy to local anesthetics
* local infection at the site of needle puncture
* parotitis
* serious liver disease
* use of antiarrhythmics group III (eg amiodarone)
* anticoagulant or antithrombotic drugs
* lactation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Time without pain | 26 weeks
  Patients will report to the investigator when pain starts to rise - and the amount of time form the procedure to the reporting will be recorded

SECONDARY OUTCOMES:
Trend of pain level | Pain level at three time points: 1 month, 3 months and 6 months after the procedure
  Pain will be graded according to visual analogue scale, 0 meaning no pain, 10 meaning the worse pain possible
Pain level when anesthesia is applied | Immediately after the procedure
  Pain will be graded according to visual analogue scale, 0 meaning no pain, 10 meaning the worse pain possible
Time to sart of the action of the block | Immediately after the procedure
  Time from the procedure till the pain is reduced, in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Monika Kocman Panic, Principal Investigator — Varazdin General Hospital
Locations (1):
- Varazdin General Hospital, Varaždin, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moore D, Chong MS, Shetty A, Zakrzewska JM. A systematic review of rescue analgesic strategies in acute exacerbations of primary trigeminal neuralgia. Br J Anaesth. 2019 Aug;123(2):e385-e396. doi: 10.1016/j.bja.2019.05.026. Epub 2019 Jun 15. PMID 31208761
- [Background] Al-Quliti KW. Update on neuropathic pain treatment for trigeminal neuralgia. The pharmacological and surgical options. Neurosciences (Riyadh). 2015 Apr;20(2):107-14. doi: 10.17712/nsj.2015.2.20140501. PMID 25864062
- [Background] Maarbjerg S, Di Stefano G, Bendtsen L, Cruccu G. Trigeminal neuralgia - diagnosis and treatment. Cephalalgia. 2017 Jun;37(7):648-657. doi: 10.1177/0333102416687280. Epub 2017 Jan 11. PMID 28076964
- [Background] Lee JY, Lee GH, Yi SH, Sim WS, Kim BW, Park HJ. Non-Surgical Treatments of Trigeminal Neuralgia from the Perspective of a Pain Physician: A Narrative Review. Biomedicines. 2023 Aug 21;11(8):2315. doi: 10.3390/biomedicines11082315. PMID 37626811
- [Background] Allam AE, Khalil AAF, Eltawab BA, Wu WT, Chang KV. Ultrasound-Guided Intervention for Treatment of Trigeminal Neuralgia: An Updated Review of Anatomy and Techniques. Pain Res Manag. 2018 Apr 2;2018:5480728. doi: 10.1155/2018/5480728. eCollection 2018. PMID 29808105
- [Background] Seo HJ, Park CK, Choi MK, Ryu J, Park BJ. Clinical Outcome of Percutaneous Trigeminal Nerve Block in Elderly Patients in Outpatient Clinics. J Korean Neurosurg Soc. 2020 Nov;63(6):814-820. doi: 10.3340/jkns.2020.0139. Epub 2020 Oct 27. PMID 33105531
- [Background] Love S, Coakham HB. Trigeminal neuralgia: pathology and pathogenesis. Brain. 2001 Dec;124(Pt 12):2347-60. doi: 10.1093/brain/124.12.2347. PMID 11701590
- [Background] Balta S, Koknel Talu G. Clinical effectiveness of peripheral nerve blocks with lidocaine and corticosteroid in patients with trigeminal neuralgia. Agri. 2021 Oct;33(4):237-242. doi: 10.14744/agri.2021.26032. PMID 34671954
- [Background] Ertilav E, Aydin ON. Evaluation of the effectiveness duration of peripheral blocks applied with high concentration local anesthetic and steroid in trigeminal neuralgia. Agri. 2022 Oct;34(4):264-271. doi: 10.14744/agri.2021.77854. PMID 36300746
- [Background] Kumar A, Sinha C, Kumar A, Kumari P, Mukul SK. Ultrasound-guided trigeminal nerve block and its comparison with conventional analgesics in patients undergoing faciomaxillary surgery: Randomised control trial. Indian J Anaesth. 2018 Nov;62(11):871-875. doi: 10.4103/ija.IJA_256_18. PMID 30532323
- [Background] Gunes A, Bulut E, Akgoz A, Mocan B, Gocmen R, Oguz KK. Trigeminal nerve and pathologies in magnetic resonance imaging - a pictorial review. Pol J Radiol. 2018 Jun 16;83:e289-e296. doi: 10.5114/pjr.2018.76921. eCollection 2018. PMID 30627249
- [Background] Jacques N, Karoutsos S, Marais L, Nathan-Denizot N. Quality of life after trigeminal nerve block in refractory trigeminal neuralgia: A retrospective cohort study and literature review. J Int Med Res. 2022 Oct;50(10):3000605221132027. doi: 10.1177/03000605221132027. PMID 36281027